CLINICAL TRIAL: NCT02814708
Title: Phase 2 Clinical Trial of the BioMed rTSST-1 Variant Vaccine in Healthy Adults
Brief Title: Clinical Trial of the BioMed rTSST-1 Variant Vaccine in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biomedizinische Forschungs gmbH (Industry)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BioMed 0515
Record Dates: First submitted 2016-06-21; First posted 2016-06-28 (Estimated); Results first posted 2021-12-13 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Toxic Shock Syndrome
Keywords: Sepsis; Vaccination
MeSH Terms: conditions — Shock, Septic; Sepsis

STUDY DESIGN:
Intervention Model Description: Two different doses of rTSST-1 Variant Vaccine were tested in different administrational schedules. These were: a comparison of 10µg versus 100µg rTSST-1 Variant Vaccine administered one, two, or three times.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Dose Group 1 (Experimental): rTSST-1 Variant Candidate Vaccine 10µg Number of Immunizations: 1
  Interventions: Biological: rTSST-1v
- Dose Group 2 (Experimental): rTSST-1 Variant Candidate Vaccine 10µg Number of Immunizations: 2
  Interventions: Biological: rTSST-1v
- Dose Group 3 (Experimental): rTSST-1 Variant Candidate Vaccine 10µg Number of Immunizations: 3
  Interventions: Biological: rTSST-1v
- Dose Group 4 (Experimental): rTSST-1 Variant Candidate Vaccine 100µg Number of Immunizations: 1
  Interventions: Biological: rTSST-1v
- Dose Group 5 (Experimental): rTSST-1 Variant Candidate Vaccine 100µg Number of Immunizations: 2
  Interventions: Biological: rTSST-1v
- Dose Group 6 (Experimental): rTSST-1 Variant Candidate Vaccine 100 µg Number of Immunizations: 3
  Interventions: Biological: rTSST-1v
- Dose Group 7 (Placebo Comparator): Al(OH)3 Adjuvant, 1mg Number of Immunizations: 3
  Interventions: Biological: rTSST-1v

INTERVENTIONS:
Biological: rTSST-1v — Each subject of a total of seven groups will receive three injections (first injection day 0; second injection 3 months ± 4 weeks after the first, third injection 6 months ± 4 weeks after the second) of one of two different doses of Vaccine or Adjuvant, each group comprising 20 subjects. Subjects will be controlled 24 h post vaccination. Follow-up will last 18 months on the average, with visits every three months (± 2 weeks). Response to treatment is defined by seroconversion from a TSST-1 binding Ab titer of < 20 to > 40 or a 4-fold increase in TSST-1 binding Ab titer .

SUMMARY:
Toxic Shock Syndrome (TSS) is a severe condition with high morbidity and mortality from the hosts overwhelming inflammatory response and cytokine storm. Staphylococcal superantigen toxins are the main causative agents. Toxic shock syndrome toxin (TSST-1) being responsible for almost all of menstruation associated and more than 50% of all other cases. There is no specific therapy.

The aim of this study is to extend the safety and tolerability of two doses of the BioMed recombinant toxic shock syndrome toxin (rTSST-1) Variant Vaccine after one to three vaccinations in healthy adults. The second aim of the study is to measure immunogenicity and persistence of antibodies which produced in response to treatment with the BioMed rTSST-1 Variant Vaccine over a period of 12 months. These antibodies are expected to be important in prevention and mitigation of the diseases. 140 healthy adults, male and female, age 18-64 years will be assigned to 7 groups comprising two doses of the vaccine or adjuvant at the Department of Clinical Pharmacology of the Medical University of Vienna. The patients will be monitored for vital signs, hematology, clinical chemistry, and antibodies against TSST-1. Immunization will be repeated 3 months after the first with the same dose and 6 months after the second immunization in the respective groups.

Antibodies will be determined through monitoring TSST-1 binding antibodies as assessed through ELISA and neutralizing antibodies (exploratory endpoint) as assessed by inhibition of T cell activation (3H Thymidine incorporation; ≥ 50%).

DETAILED DESCRIPTION:
The BioMed rTSST-1 Variant Vaccine has been developed by Biomedizinische ForschungsgmbH as one component of a polyvalent staphylococcal vaccine for the prevention of toxic shock and hyperimmunization of donors for the production of TSST-1 immunoglobulin.

This is a prospective, randomized, parallel control, phase 2 study of extended safety, local tolerance, immunogenicity, and TSST-1 antibody persistence in healthy adults, who have been vaccinated with one, two or three doses of the BioMed rTSST1 Variant Vaccine compared to adjuvant.

Over a period of 60 days prior to entry into the study, 145 male and female subjects 18 - 64 years in age will be screened for eligibility. Screening criteria will include physical examination, medical history, pregnancy/ adequate contraception in females, HIV Ab, hepatitis C virus antibodies (HCV Ab), hepatitis B antigen (HBs Ag) and TSST-1 Ab. 140 qualified subjects will be entered into the study.

Group 1 will receive 10 µg of rTSST-1 Variant Vaccine and two administrations of Adjuvant; Group 2 will receive the same dose of Vaccine twice and one dose of Adjuvant; and Group 3 will be injected the 10 µg of the Vaccine three times. Groups 4 to 6 will be given 100 µg of Vaccine following the same schedule. Group 7 will receive Al(OH3) adjuvant three times.

Prior to, and 24 h (+3 h) after each vaccination, the subjects will be examined for vital signs. Blood will be drawn for hematology, clinical chemistry tests, and C-reactive protein. Local reactions and adverse events will be assessed in all post vaccination visits.

The subjects will be followed up for a period of 3 months (± 2 weeks) or optionally 18 months (± 12 weeks) if they decide to take part in the long-term follow-up, during which they will return to the clinic every three months (± 2 weeks). Tests performed will include vital signs, local reactions, clinical chemistry, C-reactive protein. Adverse events will be recorded.

Binding and neutralizing TSST-1 antibodies will be determined prior to each vaccination and every three months during the treatment and follow-up periods.

Each participant will be in the study for 12 to 14, or optionally 24 months, if they decide to take part in the long-term follow-up.

Immunogenicity is defined by seroconversion from a TSST-1 Ab titer of < 20 to > 40 or a 4-fold increase in TSST-1 Ab titer. Neutralization will be defined as a three-fold increase of neutralization titer.

ELIGIBILITY:
Inclusion Criteria:

* males or females aged 18-64 years
* signed informed consent
* physical exam: no abnormal findings unless considered irrelevant by the investigator
* uneventful medical history
* Females with childbearing potential: adequate contraception

Exclusion Criteria:

* females with childbearing potential: pregnancy, lactation or unreliable contraception
* positive HIV Ab and/or positive HCV Ab and/or positive HBsAG signs and symptoms of autoimmunity
* TSST-1 Ab titer > 1:1000
* current or recent (< 1 month) immunosuppressive therapy with corticosteroids or immunomodulators

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2016-05; Primary Completion 2020-05 (Actual); Study Completion 2021-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha M Eibl, MD, Study Director — Biomedizinische Forschungsgmbh; Bernd Jilma, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna Department of Clinical Pharmacology, Vienna, Austria

REFERENCES:
- [Result] Schwameis M, Roppenser B, Firbas C, Gruener CS, Model N, Stich N, Roetzer A, Buchtele N, Jilma B, Eibl MM. Safety, tolerability, and immunogenicity of a recombinant toxic shock syndrome toxin (rTSST)-1 variant vaccine: a randomised, double-blind, adjuvant-controlled, dose escalation first-in-man trial. Lancet Infect Dis. 2016 Sep;16(9):1036-1044. doi: 10.1016/S1473-3099(16)30115-3. Epub 2016 Jun 10. PMID 27296693
- [Derived] Schoergenhofer C, Gelbenegger G, Hasanacevic D, Schoner L, Steiner MM, Firbas C, Buchtele N, Derhaschnig U, Tanzmann A, Model N, Larcher-Senn J, Drost M, Eibl MM, Roetzer A, Jilma B. A randomized, double-blind study on the safety and immunogenicity of rTSST-1 variant vaccine: phase 2 results. EClinicalMedicine. 2024 Jan 5;67:102404. doi: 10.1016/j.eclinm.2023.102404. eCollection 2024 Jan. PMID 38274114

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Dose Group 4 | Dose Group 5 | Dose Group 6 | Dose Group 7
Started | 20 | 20 | 20 | 20 | 20 | 20 | 20
Completed | 18 | 17 | 19 | 20 | 17 | 16 | 19
Not Completed | 2 | 3 | 1 | 0 | 3 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Dose Group 4 | Dose Group 5 | Dose Group 6 | Dose Group 7 | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 140
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (11.3) | 31.3 (11.9) | 29.2 (9.8) | 30.2 (8.5) | 31.2 (12.1) | 36.6 (11.8) | 34.2 (12.5) | 31.9 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 8 | 5 | 10 | 5 | 6 | 49
  Male | 14 | 11 | 12 | 15 | 10 | 15 | 14 | 91
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 20 | 20 | 19 | 20 | 20 | 19 | 20 | 138
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Austria | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 140

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants (Percentage) With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment
Time Frame: 12 months and 18 months follow up
Population: any suspected related systemic AE
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Dose Group 4 | Dose Group 5 | Dose Group 6 | Dose Group 7
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 20
Participants | 9 | 11 | 11 | 12 | 10 | 13 | 10

2. Secondary Outcome: Number of Participants With a Fold Increase of ELISA IgG Against rTSST-1
Description: Fold increase of antibody titer against rTSST-1 ELISA from prevaccination titer. Response to treatment is defined by seroconversion from a TSST-1 binding Ab titer of < 20 to > 40 or a 4-fold increase in TSST-1 binding Ab titer. Comparison with placebo comparator recipients.
Time Frame: 12 months and 18 months follow up
Population: per protocol population included in calculation analysed over time by treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Dose Group 4 | Dose Group 5 | Dose Group 6 | Dose Group 7
Number analyzed (Participants) | 18 | 17 | 19 | 20 | 17 | 16 | 19
Participants
  12 months | 13 | 15 | 17 | 17 | 13 | 15 | 0
  18 months | 10 | 12 | 13 | 14 | 12 | 12 | 0

ADVERSE EVENTS:
Time Frame: 27 months
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Dose Group 4 | Dose Group 5 | Dose Group 6 | Dose Group 7
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20 | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20 | 1/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 13/20 | 16/20 | 14/20 | 17/20 | 16/20 | 19/20 | 14/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Group 1 (N=20) | Dose Group 2 (N=20) | Dose Group 3 (N=20) | Dose Group 4 (N=20) | Dose Group 5 (N=20) | Dose Group 6 (N=20) | Dose Group 7 (N=20)
anaphylactic reaction (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Group 1 (N=20) | Dose Group 2 (N=20) | Dose Group 3 (N=20) | Dose Group 4 (N=20) | Dose Group 5 (N=20) | Dose Group 6 (N=20) | Dose Group 7 (N=20)
mild to moderate AE (General disorders) | 13 (39) | 16 (29) | 14 (26) | 17 (53) | 16 (39) | 19 (40) | 14 (50)
Nervos system disorders (Nervous system disorders) | 7 (25) | 10 (26) | 9 (29) | 15 (81) | 11 (30) | 10 (21) | 10 (42)
Headache (Nervous system disorders) | 6 (24) | 9 (25) | 8 (27) | 13 (75) | 11 (30) | 10 (21) | 9 (40)
General disorders and administration site conditions (General disorders) | 8 (23) | 11 (18) | 8 (15) | 13 (33) | 9 (23) | 10 (21) | 9 (24)
Fatigue (General disorders) | 6 (18) | 7 (10) | 4 (8) | 8 (15) | 5 (9) | 8 (10) | 8 (16)
Influenza-like illness (General disorders) | 2 (4) | 6 (7) | 3 (6) | 8 (12) | 6 (12) | 8 (9) | 4 (6)
Infections and infestations (Infections and infestations) | 12 (19) | 11 (25) | 12 (22) | 10 (18) | 9 (13) | 9 (20) | 10 (21)
Nasopharyngitis (Infections and infestations) | 5 (7) | 10 (18) | 6 (9) | 5 (6) | 7 (10) | 9 (16) | 6 (10)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 7 (9) | 8 (10) | 5 (7) | 11 (17) | 12 (19) | 8 (16) | 6 (9)
Gastrointestinal disorders (Gastrointestinal disorders) | 6 (6) | 7 (13) | 5 (10) | 8 (18) | 2 (2) | 5 (9) | 4 (8)
Nausea (Gastrointestinal disorders) | 2 (2) | 5 (6) | 4 (6) | 5 (10) | 1 (1) | 3 (4) | 3 (4)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 4 (4) | 3 (4) | 1 (1) | 4 (4) | 6 (8) | 3 (5) | 4 (4)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 4 (4) | 4 (5) | 6 (11) | 3 (3) | 2 (2)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 5 (6) | 4 (5) | 5 (5) | 0 (0) | 1 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 4 (4) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 5 (11) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 4 (10) | 0 (0)
Surgical and medical procedures (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (5) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (5) | 4 (4) | 6 (6) | 6 (9) | 5 (9) | 5 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (5) | 1 (1) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-20): https://cdn.clinicaltrials.gov/large-docs/08/NCT02814708/Prot_SAP_000.pdf